CLINICAL TRIAL: NCT05474235
Title: Clinical & Genetic Studies in ALS and Other Neurodegenerative Motor Neuron Disorders
Brief Title: Studies in Amyotrophic Lateral Sclerosis (ALS) and Other Neurodegenerative Motor Neuron Disorders
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Bjorn E. Oskarsson, Principal Investigator, Mayo Clinic
Other Study IDs: 07-005711; 5P01NS084974 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-26 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ALS or Suspected ALS Patient: Subjects with clinical diagnosis of possible, laboratory-supported probable, probable or definite, ALS or diagnosis of a neurodegenerative disorder with evidence of ALS plus extramotor features or a blood relative (first, second or third degree) with history of ALS or neurodegenerative disorder with evidence of ALS plus extramotor features.
- Blood Relative of ALS Patient: Subjects with family history (first, second or third degree blood relative) of ALS or other motor neuron disease.
- Healthy Control: Subjects with no personal or family history (first, second or third degree blood relative) of ALS or other motor neuron disease

SUMMARY:
The purpose of this study is to collect, from patients with sporadic and familial ALS and their family members, clinical data and blood samples for extraction of DNA, RNA, preparation of lymphocytes, plasma and serum to establish a repository for future investigations of genetic contributions to ALS pathogenesis. Blood samples for DNA extraction also would be collected from control subjects with no personal or family history of ALS phenotypes.

ELIGIBILITY:
Inclusion Criteria

ALS or Suspected ALS Patient

* Clinical diagnosis of possible, laboratory-supported probable, probable or definite ALS according to modified EL Escorial criteria, suspected ALS according to original El Escorial criteria, or diagnosis of a neurodegenerative disorder with evidence of ALS plus extramotor features; OR
* Blood relative (first, second or third degree) with history of ALS or neurodegenerative disorder with evidence of ALS plus extramotor features; OR:

  * A clinical suspicion or referral for ALS;
  * > 18 years of age;
  * Willing and able to give signed informed consent or assent that has been approved by the Institutional Review Board (IRB).

Blood Relative of ALS Patient

* Family history (first, second or third degree blood relative) of ALS or other motor neuron disease;
* > 18 years of age;
* Willing and able to give signed informed consent that has been approved by the Institutional Review Board (IRB).

Healthy Control

* No personal or family history (first, second or third degree blood relative) of ALS or other motor neuron disease;
* > 18 years of age;
* No personal history of other neurodegenerative disease (i.e., Alzheimer disease, Parkinson disease);
* Willing and able to give signed informed consent that has been approved by the Institutional Review Board (IRB).

Exclusion Criteria:

ALS or Suspected Patient • Limited mental capacity rendering the subject unable to provide written informed consent or assent or comply with standard phlebotomy procedures.

Blood Relative of ALS Patient

• Limited mental capacity rendering the subject unable to provide written informed consent or comply with standard phlebotomy procedures.

Healthy Control Subject

* Personal or family history of dementia or other neurodegenerative disease (Parkinson disease, Alzheimer disease, etc.);
* Limited mental capacity rendering the subject unable to provide written informed consent or comply with standard phlebotomy procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible subjects with ALS or suspected ALS or family history of ALS will be identified from patients seen in the Department of Neurology at Mayo Clinic Jacksonville. Inclusion criteria include standardized diagnostic criteria for ALS as used in ALS therapeutic trials and patients with clinically suspected ALS.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2007-12 (Actual); Primary Completion 2038-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Blood Collection | 50 years
  Total number of blood samples collected

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Oskarsson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No